CLINICAL TRIAL: NCT04150848
Title: A Biobehavioral Intervention for Young Men With Testicular Cancer: A Pilot Study
Brief Title: A Biobehavioral Intervention for Young Men With Testicular Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Irvine (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-4676
Record Dates: First submitted 2019-10-24; First posted 2019-11-05 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Testis Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Focused Emotion-Regulation Therapy (GET) (Experimental): GET is a 6-session intervention delivered over 8 weeks to enhance self-regulation through improved goal navigation skills, improved sense of meaning and purpose, and better ability to regulate specific emotional responses. GET has an emphasis on goal navigation skill building. This includes work on goal setting with a focus on assessing progress toward achieving specific, realistic, and measurable goals. Emotion regulation components include basic cognitive restructuring skills, cognitive distancing, and coping efficacy skills (matching the correct coping skill to specific circumstances).
  Interventions: Behavioral: Goal-Focused Emotion Regulation Therapy (GET)
- Individual Supportive Psychotherapy (ISP) (Active Comparator): ISP includes 6-sessions of individual supportive psychotherapy and includes components of genuineness, unconditional positive regard, and empathic understanding through reassurance, explanation, guidance, suggestion, encouragement, affecting changes in patient's environment, and permission for catharsis. ISP emphasizes maintaining focus on the cancer experience, supporting participants in the "here and now," fostering expression of emotion and discussion of difficult topics, and creating a sense of being understood.
  Interventions: Behavioral: Individual Supportive Psychotherapy (ISP)

INTERVENTIONS:
Behavioral: Goal-Focused Emotion Regulation Therapy (GET) — Six sessions delivered individually over 8 weeks
  Arms: Goal Focused Emotion-Regulation Therapy (GET)
Behavioral: Individual Supportive Psychotherapy (ISP) — Six sessions delivered individually over 8 weeks
  Arms: Individual Supportive Psychotherapy (ISP)

SUMMARY:
This study is a randomized controlled biobehavioral pilot trial designed to investigate the feasibility and preliminary efficacy of a novel intervention, Goal-focused Emotion-Regulation Therapy (GET) aimed at improving distress symptoms, emotion regulation, goal navigation skills, and stress-sensitive biomarkers in young adult testicular cancer patients.

Participants will be randomized to receive six sessions of GET or Individual Supportive Therapy (ISP) delivered over eight weeks. In addition to indicators of intervention feasibility, the investigators will measure primary (depressive and anxiety symptoms) and secondary (emotion regulation and goal navigation skills, career confusion) psychological outcomes prior to (T0), immediately after (T1) and twelve weeks after intervention at T2. Additionally, identified biomarkers will be measured at baseline and at T2.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 39 years at the time of consent
* confirmed diagnosis of testis cancer (any stage)
* completed chemotherapy for testis cancer within 2 years prior to consent
* fluency in English (per self-report)
* sub-optimal self-regulation as evidenced by a score of 1.8 or below on the Goal Navigation Scale or a score of 4 or greater on the Distress Thermometer (DT)

Exclusion Criteria:

* lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder (per self-report)
* active suicide plan
* disorder that compromises comprehension of assessments or informed consent information
* self-reported medical condition or medication use known to confound measures of systemic inflammation
* daily smoking

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Change from Baseline (T0) at 12-weeks Post-Intervention (T2)
  The HADS was developed to assess anxiety and depression in medical patients. It purposefully excluded somatic symptoms (e.g., sleep disturbance) to reduce confounding psychological symptoms with disease or treatment. The HADS has become a "benchmark" measure of anxiety and depression among diverse clinical and nonclinical hospital populations, including individuals diagnosed with cancer. The HADS is a 14-item self-administered questionnaire, with 7 items assigned to each the HADS-Anxiety and HADS-Depression subscales. Each item is rated on a 4-point response scale (from 0 to 3). Subscale scores are typically categorized to indicate the level of anxiety or depression experienced where scores of less than 8 are categorized as normal, scores of 8-10 as borderline, and scores of 11-21 as clinical. A number of psychometric studies have established the scale's strengths, including its brevity, reliability, and validity and availability of comparison scores across different populations.
Change in Systemic Pro-inflammatory Cytokine Levels (IL-6, IL-1ra, CRP, sTNFαRII) | Change from Baseline (T0) at intrervention completion, an average of 8 weeks
  The investigators will focus on four biomarkers, IIL-6, IL-1ra, CRP, sTNFαRII, that indicate systemic inflammation and are associated with distress symptoms and emotion regulation. Levels will be assessed from plasma. Cytokine levels will be determined by immunosorbent assay (ELISA) according to assay manufacturer's protocols. All samples will be run in duplicate, and assays will be repeated on two separate days; intra-assay and interassay mean levels will be used in all analyses.
Change in Salivary Diurnal Cortisol Slope and Daily Output | Change from Baseline (T0) at intrervention completion, an average of 8 weeks
  Diurnal rhythm in salivary cortisol will be measured over three days at each assessment. Participants will collect saliva samples in their natural environment upon awakening, 30 minutes later, 8 hours later, and at bedtime. Participants will complete a diary to assess relevant health behaviors (e.g., caffeine, tobacco, alcohol consumption; physical activity, sleep) as well as daily stress. They will be instructed to avoid brushing their teeth, eating, or drinking within 20 minutes before sampling. Participants will keep samples refrigerated prior to returning them to the research laboratory and returned salivettes will be stored in a -20-degree Celsius freezer until analyzed. After data collection is complete, salivary cortisol will be analyzed with a time-resolved fluorescence immunoassay at the IISBR laboratory at UC Irvine. Several indices will be computed including diurnal slope, area under the daily curve, cortisol awakening response, and total daily cortisol output.

SECONDARY OUTCOMES:
Change in Emotion Regulation Questionnaire (ERQ) Scale Scores | Change from Baseline (T0) at 12-weeks Post-Intervention (T2)
  Emotion regulation skills will be measured by the Emotion Regulation Questionnaire (ERQ). The ERQ is a widely used 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The ERQ is widely used in the context of clinical treatment trials and has well established validity, reliability, and factor structure (Goldin, Manber-Ball, Werner, Heimberg, & Gross, 2009; Gross & John, 2003).
Change in Cancer Assessment for Young Adults (CAYA-T) - Goal Navigation Score | Change from Baseline (T0) at 12-weeks Post-Intervention (T2)
  Goal navigation capacity includes elements of goal setting, goal clarification, goal adjustment, and goal initiation. It will be measured by the Goal Navigation subscale of the Cancer Assessment for Young Adults -Testicular (CAYA-T) (Hoyt et al., 2013). The scale is composed of five items (e.g., "I am able to identify goals in my life", "I know what steps to take to make progress toward my goals", and "I am able to redirect my energy when I feel my life isn't going in the right direction"). Participants indicate how often each item is true of them over the past 7 days on a 3-point response scale ranging from 0 (None of the time) to 2 (Much or most of the time). Criterion, construct, and procedural validity have been established with young adult testicular cancer survivors.
Change in Career Thoughts Inventory (CTI) Global Score | Change from Baseline (T0) at 12-weeks Post-Intervention (T2)
  The CTI (Sampson et al., 1996) is a 48-item self-administered instrument that measures an individual's level of dysfunctional thinking in career decision-making and career problem-solving. The CTI is normed on adults and broadly used in the context of I/O Psychology. Items are rated on a 4-point Likert scale ranging from 0 (strongly disagree) to 3 (strongly agree). CTI total score provides information about an individual's overall level of dysfunctional career thoughts, However, the CTI has three subscales: Decision-Making Confusion (difficulties with initiating or sustaining a career choice), Commitment Anxiety (difficulties with making a commitment to a career choice), and External Conflict (difficulties with balancing one's ideas with the ideas from others). The CTI has sound evidence for its content, construct, and criterion-related validity (Peila-Shuster & Feller, 2013; Sampson et al., 1996).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request with permission of the investigation team.

REFERENCES:
- [Derived] Hoyt MA, Wang AW, Ceja RC, Cheavens JS, Daneshvar MA, Feldman DR, Funt SA, Nelson CJ. Goal-Focused Emotion-Regulation Therapy (GET) in Young Adult Testicular Cancer Survivors: A Randomized Pilot Study. Ann Behav Med. 2023 Aug 21;57(9):777-786. doi: 10.1093/abm/kaad010. PMID 37078969
- [Derived] Hoyt MA, Wang AW, Ryan SJ, Breen EC, Cheavens JS, Nelson CJ. Goal-Focused Emotion-Regulation Therapy (GET) for young adult survivors of testicular cancer: a pilot randomized controlled trial of a biobehavioral intervention protocol. Trials. 2020 Apr 14;21(1):325. doi: 10.1186/s13063-020-04242-0. PMID 32290859